CLINICAL TRIAL: NCT06740123
Title: Clinical, Radiological, and Biochemical Evaluation of Adjunctive Hydrogel Application in the Non-Surgical Treatment of Peri-implantitis and Periodontitis
Brief Title: Evaluation of Hydrogel Application in the Treatment of Periodontitis and Peri-implantitis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Berceste Guler, Associate Professor Dr., Kutahya Health Sciences University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023-15/01
Record Dates: First submitted 2024-11-27; First posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-11

CONDITIONS: Periodontal Disease Stage 2; Peri-Implantitis and Peri-implant Mucositis; Periodontal Regeneration
Keywords: Periodontitis; Peri-implantitis; Hydrogel; non-surgical periodontal treatment
MeSH Terms: conditions — Periodontal Diseases; Peri-Implantitis; Periodontitis

STUDY DESIGN:
Intervention Model Description: A total of 30 patients, including 15 systemically healthy patients older than 18 years of age, with Stage 2 periodontitis and periodontal/peri-implant pockets between 5-8 mm on the contralateral side, who applied to Kütahya Health Sciences University, Faculty of Dentistry, Department of Periodontology, will be included in the study. Patients with periodontal/peri-implant pockets will be evaluated in a total of four groups after non-surgical periodontal treatment, two different groups, one side of the patients will be the test group and the other side will be the control group. All patients will be randomly allocated to the study groups using the sealed envelope method.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Periodontal pocket (Test group) (Experimental): To be treated with non-surgical periodontal treatment and intra-pocket H42 hydrogel application.
  Interventions: Procedure: Non-surgical periodontal treatment and application of H42® hydrogel to the periodontal pocket
- Periodontal pocket (Control group) (Experimental): To be treated with non-surgical periodontal treatment only
  Interventions: Procedure: Nonsurgical periodontal treatment of periodontal pocket
- Peri-implant pocket (Test group) (Experimental): Will be treated with non-surgical periodontal treatment and intra-pocket H42 hydrogel application.
  Interventions: Procedure: Nonsurgical periodontal treatment and application of H42® hydrogel to the peri-implant pocket
- Peri-implant pocket (Control group) (Experimental): will be treated with non-surgical periodontal treatment only
  Interventions: Procedure: Nonsurgical periodontal treatment of peri-implant pocket

INTERVENTIONS:
Procedure: Nonsurgical periodontal treatment and application of H42® hydrogel to the peri-implant pocket — Firstly, after appropriate oral hygiene training, full mouth supragingival scaling will be performed using an ultrasonic device (EMS Piezon ultrasonic system, EMS Electro Medical Systems, Switzerland). Non-surgical periodontal treatment will be completed after subgingival curettage of peri-implant pocket areas between 5-8 mm in the contralateral quadrant. The tested site will be partially isolated and then air-dried. A bent, blunt-tipped needle syringe will be used to inject the H42® hydrogel into the pocket, ensuring that the tip reaches the deepest point of the pocket. Once the gel is visible at the gingival margin, the needle will be gently removed from the pocket. After approximately 0.1 mL of gel has been applied, excess gel will be removed with a sterile gauze swab to prevent any spreading effect or possible systemic effect. After application of the H42 hydrogel, the area will be kept dry for 5 minutes to ensure optimum adhesion of H42 to the pocket tissue.
  Arms: Peri-implant pocket (Test group)
Procedure: Nonsurgical periodontal treatment of periodontal pocket — Systemic and dental anamnesis will be taken from all patients. Firstly, after appropriate oral hygiene education, full mouth supragingival scaling will be performed using an ultrasonic device (EMS Piezon ultrasonic system, EMS Electro Medical Systems, Switzerland). Non-surgical periodontal treatment will be completed after subgingival curettage of periodontal pocket areas between 5-8 mm in the contralateral quadrant.
  Arms: Periodontal pocket (Control group)
Procedure: Non-surgical periodontal treatment and application of H42® hydrogel to the periodontal pocket — Firstly, after appropriate oral hygiene training, full mouth supragingival scaling will be performed using an ultrasonic device (EMS Piezon ultrasonic system, EMS Electro Medical Systems, Switzerland). Non-surgical periodontal treatment will be completed after subgingival curettage of periodontal pocket areas between 5-8 mm in the contralateral quadrant. The tested site will be partially isolated and then air-dried. A bent, blunt-tipped needle syringe will be used to inject the H42® hydrogel into the pocket, ensuring that the tip reaches the deepest point of the pocket. Once the gel is visible at the gingival margin, the needle will be gently removed from the pocket. After approximately 0.1 mL of gel has been applied, excess gel will be removed with a sterile gauze swab to prevent any spreading effect or possible systemic effect. After application of the H42 hydrogel, the area will be kept dry for 5 minutes to ensure optimum adhesion of H42 to the pocket tissue.
  Arms: Periodontal pocket (Test group)
Procedure: Nonsurgical periodontal treatment of peri-implant pocket — Systemic and dental anamnesis will be taken from all patients. Firstly, after appropriate oral hygiene education, full mouth supragingival scaling will be performed using an ultrasonic device (EMS Piezon ultrasonic system, EMS Electro Medical Systems, Switzerland). Non-surgical periodontal treatment will be completed after subgingival curettage of peri-implant pocket areas between 5-8 mm in the contralateral quadrant.
  Arms: Peri-implant pocket (Control group)

SUMMARY:
To date, systemic/local antibiotics, antimicrobials, laser application, and probiotics have been used as adjuncts to improve the outcome of non-surgical periodontal treatment for both periodontitis and peri-implantitis patients. H42® hydrogel, obtained by combining a high molecular weight hydrogel with type I collagen, is a collagen paste for regenerating periodontal/peri-implant pockets caused by periodontitis/peri-implantitis. This study aimed to clinically, biochemically, and radiologically evaluate the effect and reliability of hydrogel application into the pocket in addition to non-surgical periodontal treatment in the treatment of periodontal and peri-implant pockets.

Fifteen patients with stage 2 periodontitis, each with 30 teeth and 30 implants with 5-8 mm pocket depth in the contralateral quadrants, and a total of 30 patients, will be equally divided into two groups. The test group will receive non-surgical periodontal treatment followed by H42 hydrogel application (Hydrogel Oral- 3 syr 0.4 cc/syr), while the control group will receive only non-surgical periodontal treatment. All patients will undergo the same procedure of non-surgical periodontal treatment

DETAILED DESCRIPTION:
Periodontitis is a chronic, multifactorial, inflammatory disease associated with biofilm and characterized by the destruction of the bone supporting the tooth. Peri-implantitis is an inflammatory disease associated with inflammation of the peri-implant mucosa followed by progressive bone destruction of varying degrees, with a peri-implant pocket depth of at least 4 mm, accompanied by symptoms such as bleeding and suppuration. Peri-implantitis and periodontitis have similar microbial flora, but peri-implantitis is more complex. In periodontitis and peri-implantitis patients, adjunctive therapies are needed to support non-surgical treatment and to strengthen the immune system by suppressing periodontal pathogens. Adjunctive therapies include local and systemic antibiotics, laser applications, antimicrobials, probiotics, photodynamic therapy, host-modulating agents, enamel matrix protein, injectable platelet-rich fibrin, hyaluronic acid gel, and other medications. H42® hydrogel, obtained by combining a high molecular weight hydrogel with type I collagen; It is an applied collagen paste that helps non-surgical periodontal treatment of periodontal and peri-implant diseases with its physical, bio-chemical, and rheological properties. The plugging effect and visco-elasticity of the hydrogel limits bacterial recolonisation after the use of mechanical instruments in periodontal/peri-implant pockets and allow the regeneration of periodontal/peri-implant pockets caused by periodontitis/peri-implantitis. When the H42® hydrogel is applied to the affected area, it physically moves away from the implant site over a period of 15-30 days and does not need to be removed from the application site.

To evaluate clinically, biochemically and radiologically the effect and reliability of hydrogel application into the pocket in addition to non-surgical periodontal treatment in the treatment of periodontitis/peri-implantitis patients with periodontal/peri-implant pockets between 5-8 mm contralaterally.

A total of 30 patients, including 15 systemically healthy patients older than 18 years of age, with Stage 2 periodontitis and periodontal/peri-implant pockets between 5-8 mm on the contralateral side, who applied to Kütahya Health Sciences University, Faculty of Dentistry, Department of Periodontology, will be included in the study.

Study group periodontal pockets: Thirty teeth in 15 patients with stage 2 periodontitis with 5-8 mm pocket depth in the contralateral quadrants will be equally divided into two groups.

Group I (Test Group) (number of pockets = 15): Will be treated with nonsurgical periodontal treatment and intrapocket H42 hydrogel application.

Group II (Control Group) (number of pockets = 15): Will be treated with nonsurgical periodontal treatment only.

Study group peri-implant pockets:Thirty implants in 15 patients with stage 2 periodontitis with 5-8 mm pocket depth in the contralateral quadrants will be equally divided into two groups.

Group III (Test Group) (number of pockets = 15): Will be treated with nonsurgical periodontal treatment and intrapocket H42 hydrogel application.

Group IV (Control Group) (number of pockets = 15): Will be treated with nonsurgical periodontal treatment only.

All patients will be randomly allocated to study groups using the sealed envelope method. The test group will receive non-surgical periodontal treatment followed by H42 hydrogel application (Hydrogel Oral- 3 syr 0.4 cc/syr), while the control group will receive only non-surgical periodontal treatment. All patients will undergo the same procedure of non-surgical periodontal treatment (scaling and subgingival curettage treatment) with ultrasonic instrument (EMS Piezon ultrasonic system, EMS Electro Medical Systems, Switzerland). Non-surgical periodontal treatment will be completed after subgingival curettage of periodontal or peri-implant pocket sites between 5-8 mm in the contralateral quadrant. For the test group only, the tested site will be partially isolated and then air-dried. A bent, blunt-tipped needle syringe will be used to inject the hydrogel (H42) into the pocket, ensuring that the tip is inserted into the deepest point of the pocket. Once the gel is visible at the gingival margin, the needle will be gently removed from the pocket. After approximately 0.1 mL of gel has been applied, excess gel will be removed with a sterile gauze swab to prevent any spreading effect or possible systemic effect as a result of swallowing the gel. After application of the H42 hydrogel, the site will be kept dry for 5 minutes to ensure optimum adhesion of H42 to the pocket tissue. Patients will be advised to practice normal oral hygiene with no restrictions on dietary habits and to check for any re-infection. Periodontal clinical measurements (plaque index, gingival index, clinical attachment loss, bleeding index on probing and pocket depth) will be recorded at all implant and natural tooth sites with a pre-calibrated graduated William periodontal probe by a single clinician at baseline, 1 month, and 3 months after treatment. For biochemical evaluation, gingival crevicular fluid samples will be collected from the deepest pocket depth sites of all patients, from the test and control groups, at baseline, 1 month, and 3 months after treatment. The preferred time for collecting gingival crevicular fluid samples will be between 09:00-14:00. Gingival crevicular fluid samples will be collected from the mesial, distal, buccal and lingual surfaces of teeth or implants using standard-sized paper strips. The areas to be sampled will be isolated and the teeth will be lightly dried. The previously prepared paper strips placed in the pockets will be advanced until resistance is felt in the sulcus and will be kept in the pocket for 30 seconds. The gingival crevicular fluid samples obtained will be analyzed for IL-6, Prostaglandin E2 and IL-1 beta and TNF-alpha by ELISA. Periodontal radiographic evaluation will be performed on periapical x-rays taken with parallel technique from the relevant implant and tooth area before treatment and at 3-month follow-up. In addition, a 3D cone beam computed tomography image will be obtained to understand the shape of the bone destruction defect around the relevant tooth and implant and to measure the amount of bone filling 6 months after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. be over 18 years old
2. The patient does not have any systemic disease
3. Patients with a probed pocket depth of 5-8 mm in at least one tooth in the opposite quadrant
4. According to the 2017 World Workshop on Classification of Periodontal and Peri-Implant Diseases and Conditions, patients of both sexes, aged 25-50 years, diagnosed with stage 2, grade B periodontitis
5. Patients with clinical loss of attachment of 3-4 mm, bleeding during probing and radiographic horizontal bone loss in the coronal third of the root (15-33%)
6. Clinical attachment loss of 3-4 mm in <30% of teeth associated with periodontitis
7. Patients with a radiographic bone loss/age of 0.25-1 on the tooth with the greatest bone loss in the degree of periodontitis
8. Patients without anti-inflammatory drug use in the last 2 months
9. Patients who have not received antibiotic treatment in the last 6 months

Exclusion Criteria:

1. Any systemic disease that may adversely affect the results of treatment (receiving radiotherapy and chemotherapy, systemic bisphosphonate, and corticosteroid use) to be found
2. To have undergone a surgical operation in the same region within the last 3 months
3. Smoking patients
4. Pregnancy
5. Presence of systemic conditions requiring antibiotic prophylaxis
6. Acute and untreated periodontitis
7. Patients receiving simultaneous treatment with a hyaluronic acid gel

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Periodontal or peri-implant pocket depth | 3-month follow-up of all implants and teeth
  The primary outcome was the distance between the base of the periodontal sulcus and the gingival margin measured with a standard periodontal probe at 3-month follow-up.
Proinflammatory markers | 3-month follow-up of all implants and teeth
  Gingival crevicular fluid samples are analyzed for proinflammatory markers IL-6, Prostaglandin E2 and IL-1 beta and TNF-alpha using the ELISA method at 3-months follow-up.
Marginal bone level change | 6-month follow-up of all implants and teeth
  The primary outcome was measurement of marginal bone level on periapical radiographs and cone-beam computed tomography at 6-month follow-up.

SECONDARY OUTCOMES:
Patients participating in the evaluation of a treatment may encounter both adverse and beneficial events associated with that treatment | 6-month follow-up of all implants and teeth
  Both adverse and beneficial events associated with the evaluated treatment will be systematically documented for each patient at 6 months. The change in patients' pain scores on the Numerical Rating Scale from baseline to 3 months after treatment will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Berceste Güler Ayyıldız, Assoc. Prof. Dr, Study Director — Kütahya Health Sciences University
Locations (1):
- Kütahya Health Sciences University Faculty of Dentistry, Kütahya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol
  Statistical Analysis Plan (SAP)
Supporting Information: Study Protocol, SAP
Time Frame: The work will be shared 6 months after publication.
Access Criteria: It will be shared in case the principal investigator is contacted.

REFERENCES:
- [Background] Kanjevac T, Taso E, Stefanovic V, Petkovic-Curcin A, Supic G, Markovic D, Djukic M, Djuran B, Vojvodic D, Sculean A, Rakic M. Estimating the Effects of Dental Caries and Its Restorative Treatment on Periodontal Inflammatory and Oxidative Status: A Short Controlled Longitudinal Study. Front Immunol. 2021 Sep 15;12:716359. doi: 10.3389/fimmu.2021.716359. eCollection 2021. PMID 34603290
- [Background] Zhou Y, Petpichetchian W, Kitrungrote L. Psychometric properties of pain intensity scales comparing among postoperative adult patients, elderly patients without and with mild cognitive impairment in China. Int J Nurs Stud. 2011 Apr;48(4):449-57. doi: 10.1016/j.ijnurstu.2010.08.002. PMID 20817183
- [Background] Zhou S, Miao D, Wen J, Zhang Q, Hu D, Liu N, Li J, Zhang Y, Wang K, Chen Y. Microcin C7-laden modified gelatin based biocomposite hydrogel for the treatment of periodontitis. Int J Biol Macromol. 2024 Feb;258(Pt 1):128293. doi: 10.1016/j.ijbiomac.2023.128293. Epub 2023 Nov 22. PMID 38000587
- [Background] Santos MS, Dos Santos AB, Carvalho MS. New Insights in Hydrogels for Periodontal Regeneration. J Funct Biomater. 2023 Nov 11;14(11):545. doi: 10.3390/jfb14110545. PMID 37998114
- [Background] Ivanov AA, Kuznetsova AV, Popova OP, Danilova TI, Latyshev AV, Yanushevich OO. Influence of Extracellular Matrix Components on the Differentiation of Periodontal Ligament Stem Cells in Collagen I Hydrogel. Cells. 2023 Sep 22;12(19):2335. doi: 10.3390/cells12192335. PMID 37830549
- [Background] Linares A, Sanz-Sanchez I, Dopico J, Molina A, Blanco J, Montero E. Efficacy of adjunctive measures in the non-surgical treatment of peri-implantitis: A systematic review. J Clin Periodontol. 2023 Jun;50 Suppl 26:224-243. doi: 10.1111/jcpe.13821. Epub 2023 May 4. PMID 37143407
- [Background] Ambili R, Nazimudeen NB. Adjunctive benefit of probiotic supplementation along with nonsurgical therapy for peri-implant diseases - A systematic review and meta-analysis. J Indian Soc Periodontol. 2023 Jul-Aug;27(4):352-361. doi: 10.4103/jisp.jisp_308_22. Epub 2023 Jul 1. PMID 37593565
- [Background] Altindal D, Alkan EA, Calisir M. Evaluation of the effectiveness of diode laser therapy in conjunction with nonsurgical treatment of peri-implantitis. J Periodontal Implant Sci. 2023 Oct;53(5):376-387. doi: 10.5051/jpis.2203140157. Epub 2023 Feb 3. PMID 37038829
- [Background] Mombelli A, Feloutzis A, Bragger U, Lang NP. Treatment of peri-implantitis by local delivery of tetracycline. Clinical, microbiological and radiological results. Clin Oral Implants Res. 2001 Aug;12(4):287-94. doi: 10.1034/j.1600-0501.2001.012004287.x. English, French, German. PMID 11488856
- [Background] Linares A, Pico A, Blanco C, Blanco J. Adjunctive Systemic Metronidazole to Nonsurgical Therapy of Peri-implantitis with Intrabony Defects: A Retrospective Case Series Study. Int J Oral Maxillofac Implants. 2019 Sep/Oct;34(5):1237-1245. doi: 10.11607/jomi.7343. PMID 31528867
- [Background] Estefania-Fresco R, Garcia-de-la-Fuente AM, Egana-Fernandez-Valderrama A, Bravo M, Aguirre-Zorzano LA. One-year results of a nonsurgical treatment protocol for peri-implantitis. A retrospective case series. Clin Oral Implants Res. 2019 Jul;30(7):702-712. doi: 10.1111/clr.13456. Epub 2019 Jun 1. PMID 31090974
- [Background] Daubert D, Lee E, Botto A, Eftekhar M, Palaiologou A, Kotsakis GA. Assessment of titanium release following non-surgical peri-implantitis treatment: A randomized clinical trial. J Periodontol. 2023 Sep;94(9):1122-1132. doi: 10.1002/JPER.22-0716. Epub 2023 May 2. PMID 37070363
- [Background] Schwarz F, Ramanauskaite A. It is all about peri-implant tissue health. Periodontol 2000. 2022 Feb;88(1):9-12. doi: 10.1111/prd.12407. PMID 35103327
- [Background] Renvert S, Polyzois I, Persson GR. Treatment modalities for peri-implant mucositis and peri-implantitis. Am J Dent. 2013 Dec;26(6):313-8. PMID 24640434
- [Background] Figuero E, Graziani F, Sanz I, Herrera D, Sanz M. Management of peri-implant mucositis and peri-implantitis. Periodontol 2000. 2014 Oct;66(1):255-73. doi: 10.1111/prd.12049. PMID 25123773
- [Background] Derks J, Ichioka Y, Dionigi C, Trullenque-Eriksson A, Berglundh J, Tomasi C, Graziani F. Prevention and management of peri-implant mucositis and peri-implantitis: A systematic review of outcome measures used in clinical studies in the last 10 years. J Clin Periodontol. 2023 May;50 Suppl 25:55-66. doi: 10.1111/jcpe.13608. Epub 2022 Jul 11. PMID 35246865
- [Background] Schwarz F, Derks J, Monje A, Wang HL. Peri-implantitis. J Clin Periodontol. 2018 Jun;45 Suppl 20:S246-S266. doi: 10.1111/jcpe.12954. PMID 29926484
- [Background] Dreyer H, Grischke J, Tiede C, Eberhard J, Schweitzer A, Toikkanen SE, Glockner S, Krause G, Stiesch M. Epidemiology and risk factors of peri-implantitis: A systematic review. J Periodontal Res. 2018 Oct;53(5):657-681. doi: 10.1111/jre.12562. Epub 2018 Jun 7. PMID 29882313
- [Background] Berglundh T, Armitage G, Araujo MG, Avila-Ortiz G, Blanco J, Camargo PM, Chen S, Cochran D, Derks J, Figuero E, Hammerle CHF, Heitz-Mayfield LJA, Huynh-Ba G, Iacono V, Koo KT, Lambert F, McCauley L, Quirynen M, Renvert S, Salvi GE, Schwarz F, Tarnow D, Tomasi C, Wang HL, Zitzmann N. Peri-implant diseases and conditions: Consensus report of workgroup 4 of the 2017 World Workshop on the Classification of Periodontal and Peri-Implant Diseases and Conditions. J Clin Periodontol. 2018 Jun;45 Suppl 20:S286-S291. doi: 10.1111/jcpe.12957. PMID 29926491
- [Background] Tarnow DP. Increasing Prevalence of Peri-implantitis: How Will We Manage? J Dent Res. 2016 Jan;95(1):7-8. doi: 10.1177/0022034515616557. No abstract available. PMID 26701918
- [Background] Ginesin O, Mayer Y, Gabay E, Rotenberg D, Machtei EE, Coyac BR, Bar-On Y, Zigdon-Giladi H. Revealing leukocyte populations in human peri-implantitis and periodontitis using flow cytometry. Clin Oral Investig. 2023 Sep;27(9):5499-5508. doi: 10.1007/s00784-023-05168-y. Epub 2023 Jul 25. PMID 37490117
- [Background] Lafaurie GI, Sabogal MA, Castillo DM, Rincon MV, Gomez LA, Lesmes YA, Chambrone L. Microbiome and Microbial Biofilm Profiles of Peri-Implantitis: A Systematic Review. J Periodontol. 2017 Oct;88(10):1066-1089. doi: 10.1902/jop.2017.170123. Epub 2017 Jun 19. PMID 28625077
- [Background] Turkmen M, Firatli E. The study of genetic predisposition on periodontitis and peri-implantitis. Niger J Clin Pract. 2022 Nov;25(11):1799-1804. doi: 10.4103/njcp.njcp_19_22. PMID 36412285
- [Background] Shunmuga PD, Tadepalli A, Parthasarathy H, Ponnaiyan D, Cholan PK, Ramachandran L. Clinical evaluation of the combined efficacy of injectable platelet-rich fibrin along with scaling and root planing in the non-surgical periodontal therapy of stage III and grade C periodontitis patients having type 2 diabetes mellitus: A randomized controlled trial. Clin Adv Periodontics. 2024 Sep;14(3):223-231. doi: 10.1002/cap.10266. Epub 2023 Sep 25. PMID 37749861
- [Background] Ramanauskaite E, Machiulskiene V, Dvyliene UM, Eliezer M, Sculean A. Clinical Evaluation of a Novel Combination of Sodium Hypochlorite/Amino Acid and Cross-linked Hyaluronic Acid Adjunctive to Non-surgical Periodontal Treatment: A Case Series. Oral Health Prev Dent. 2023 Aug 30;21:279-284. doi: 10.3290/j.ohpd.b4347453. PMID 37724897
- [Background] Abu-Ta'a M, Marzouka D. Enamel Matrix Derivative (EMD) as an Adjunct to Non-surgical Periodontal Therapy: A Systematic Review. Cureus. 2023 Aug 15;15(8):e43530. doi: 10.7759/cureus.43530. eCollection 2023 Aug. PMID 37719602
- [Background] El Mobadder M, Nammour S, Grzech-Lesniak K. Photodynamic Therapy with Tolonium Chloride and a Diode Laser (635 nm) in the Non-Surgical Management of Periodontitis: A Clinical Study. J Clin Med. 2023 Aug 13;12(16):5270. doi: 10.3390/jcm12165270. PMID 37629310
- [Background] Alhamoudi N, Abduljabbar T, Vohra F, Javed F. Influence of mechanical debridement with adjunct probiotic therapy on clinical status and salivary cortisol levels in patients with periodontal inflammation. Eur Rev Med Pharmacol Sci. 2023 Sep;27(18):8360-8370. doi: 10.26355/eurrev_202309_33758. PMID 37782153
- [Background] Sanz M, Herrera D, Kebschull M, Chapple I, Jepsen S, Beglundh T, Sculean A, Tonetti MS; EFP Workshop Participants and Methodological Consultants. Treatment of stage I-III periodontitis-The EFP S3 level clinical practice guideline. J Clin Periodontol. 2020 Jul;47 Suppl 22(Suppl 22):4-60. doi: 10.1111/jcpe.13290. PMID 32383274
- [Background] Herrera D, Matesanz P, Bascones-Martinez A, Sanz M. Local and systemic antimicrobial therapy in periodontics. J Evid Based Dent Pract. 2012 Sep;12(3 Suppl):50-60. doi: 10.1016/S1532-3382(12)70013-1. PMID 23040339
- [Background] Caton JG, Armitage G, Berglundh T, Chapple ILC, Jepsen S, Kornman KS, Mealey BL, Papapanou PN, Sanz M, Tonetti MS. A new classification scheme for periodontal and peri-implant diseases and conditions - Introduction and key changes from the 1999 classification. J Clin Periodontol. 2018 Jun;45 Suppl 20:S1-S8. doi: 10.1111/jcpe.12935. PMID 29926489
- [Background] Sabharwal A, Gomes-Filho IS, Stellrecht E, Scannapieco FA. Role of periodontal therapy in management of common complex systemic diseases and conditions: An update. Periodontol 2000. 2018 Oct;78(1):212-226. doi: 10.1111/prd.12226. PMID 30198128
- [Background] Mainas G, Ide M, Rizzo M, Magan-Fernandez A, Mesa F, Nibali L. Managing the Systemic Impact of Periodontitis. Medicina (Kaunas). 2022 Apr 29;58(5):621. doi: 10.3390/medicina58050621. PMID 35630038
- [Background] Zhang Y, Zhang Y, Mei Y, Zou R, Niu L, Dong S. Reactive Oxygen Species Enlightened Therapeutic Strategy for Oral and Maxillofacial Diseases-Art of Destruction and Reconstruction. Biomedicines. 2022 Nov 11;10(11):2905. doi: 10.3390/biomedicines10112905. PMID 36428473
- [Background] Papapanou PN, Sanz M, Buduneli N, Dietrich T, Feres M, Fine DH, Flemmig TF, Garcia R, Giannobile WV, Graziani F, Greenwell H, Herrera D, Kao RT, Kebschull M, Kinane DF, Kirkwood KL, Kocher T, Kornman KS, Kumar PS, Loos BG, Machtei E, Meng H, Mombelli A, Needleman I, Offenbacher S, Seymour GJ, Teles R, Tonetti MS. Periodontitis: Consensus report of workgroup 2 of the 2017 World Workshop on the Classification of Periodontal and Peri-Implant Diseases and Conditions. J Clin Periodontol. 2018 Jun;45 Suppl 20:S162-S170. doi: 10.1111/jcpe.12946. PMID 29926490